CLINICAL TRIAL: NCT04168008
Title: A Randomized Controlled Trial of Women Involved in Supporting Health (WISH), a Peer-Led Intervention to Improve Postpartum Retention in HIV Care
Brief Title: A Peer-Led Intervention to Improve Postpartum Retention in HIV Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Florence Momplaisir, MD, Assistant Professor, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 833893; 1R01MD013558 (NIH)
Record Dates: First submitted 2019-11-08; First posted 2019-11-19 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: HIV/AIDS
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants will be assigned in equal proportions to either the WISH Adherence arm or to the WISH Parenting arm
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adherence (Experimental): Women randomized to the adherence arm will attend 3 prenatal sessions and 2 postpartum sessions with a peer facilitator. Each session will be delivered on an individual basis and consist of structured educational content followed by unstructured conversation, allowing the participant to ask questions and actively engage in formulating her plan to be retained in HIV care. The goal of the prenatal sessions is to introduce the intervention, foster bonding, and address outcome expectancies and self-efficacy regarding retention in HIV care postpartum. The postpartum sessions build on outcome expectancies and self-efficacy to develop skills for Antiretroviral therapy (ART) adherence and engagement in HIV care.
  Interventions: Behavioral: WISH Adherence
- Parenting (Active Comparator): Women randomized to the parenting control arm will also attend 3 prenatal sessions and 2 postpartum sessions with a peer facilitator. The educational sessions will be focused on parenting and baby care.
  Interventions: Behavioral: WISH Parenting

INTERVENTIONS:
Behavioral: WISH Adherence — The educational sessions will consist of an adherence-centered curriculum.
  Arms: Adherence
Behavioral: WISH Parenting — The educational sessions will focus on parenting and baby care.
  Arms: Parenting

SUMMARY:
The purpose of this study is to test the efficacy of a theory-driven peer intervention for pregnant and postpartum women living HIV. The peer intervention is designed to increase self-efficacy, social support, self-regulatory behaviors, and outcome expectancy in order to improve retention in care and viral suppression postpartum. The intervention will consist of face-to-face prenatal educational sessions, starting in early third trimester, and postpartum sessions scheduled up to three months postpartum.

DETAILED DESCRIPTION:
Despite significant progress in the reduction of perinatal transmission of HIV, there has been less attention to retaining women living with HIV (WLH) in care in the postpartum period. Retention in care particularly affects black and Hispanic women as they are disproportionately affected by the HIV epidemic in the United States (U.S.). In preliminary work, the investigators used HIV surveillance data from the Philadelphia Department of Public Health to examine the HIV care continuum of 561 women, 78% of whom were black, during pregnancy and up to two years postpartum (2005-2011). Only 38% of women received HIV care within 3 months after delivery, and retention remained poor at 1 (39%) and 2 (25%) years postpartum. Poor maternal retention in care also occurs in Mississippi, Georgia, and New York, demonstrating that this break in the HIV care continuum is widespread. Retaining WLH in care positively impacts their well-being and health postpartum and for years to come, which promotes not only their health but that of their newborns. Therefore, the long-term goal of this study is to decrease HIV disparities by increasing WLH's retention in care in the postpartum period.

Presently, there are a limited number of evidence-based interventions aimed at improving retention in care for WLH. Through a critical review of research literature, the investigators found that interventions to improve retention in care have been implemented in low-resource countries, but studies in high-resource countries are lacking. In sub-Saharan Africa, the use of peers has resulted in significantly higher maternal retention and viral suppression compared to standard of care. Peers are WLH who remained engaged in HIV care postpartum, and provide education and support to WLH in the prenatal and postpartum periods. The investigators also conducted a series of qualitative interviews with WLH in the U.S. to evaluate factors contributing to poor retention in care postpartum, and to assess the acceptability and feasibility of a peer intervention in meeting women's needs. The results showed that women's primary motivation to engage in prenatal care is to keep their infant healthy, but that many of them experience significant life challenges that impede their ability to engage in care postpartum. However, they expressed great interest in receiving support from a peer to motivate sustained engagement in care postpartum.

The investigators propose to test the efficacy of a theory-driven peer intervention, based on the integrated model of health behavior. The peer intervention, Women Involved in Supporting Health (WISH), is designed to increase self-efficacy, social support, self-regulatory behaviors, and outcome expectancy in order to improve retention in care and viral suppression postpartum. The intervention will consist of three face-to-face prenatal sessions, starting in early third trimester, and two face-to-face postpartum sessions scheduled up to three months postpartum. The prenatal sessions focus on knowledge that will address barriers to outcome expectancies and self-efficacy, and the postpartum sessions build on outcome expectancy and knowledge to develop skills tailored to adherence to antiretroviral therapy and engagement in HIV care. Between the sessions, the peer and the WLH will communicate via text messages, phone calls and/or video chat. The randomized controlled trial (RCT) will take place across Center for AIDS Research sites in Philadelphia, the District of Columbia, Atlanta, and Birmingham, where HIV infection rates remain disproportionally high among black and Hispanic women. A total of 260 pregnant WLH will be randomized to either WISH adherence or an attention-matched WISH parenting control group.

The impact of this research will be the development of the first evidence-based peer intervention to address the pressing need to improve postpartum retention in HIV care and viral suppression of WLH in the U.S.

ELIGIBILITY:
Inclusion Criteria:

* 16 years and older
* a woman living with HIV in the 2nd or 3rd trimester of pregnancy
* able to provide informed consent including HIPAA authorization to access protected health information
* able to read and speak English
* having access to a cell phone

Exclusion Criteria:

* planning to relocate outside the country within the year following delivery

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2020-03-03 (Actual); Primary Completion 2025-09-08 (Actual); Study Completion 2025-09-08 (Actual)

PRIMARY OUTCOMES:
Retention in Care up to 1 year postpartum | Baseline through 1 year after delivery
  ≥1 visit with an HIV provider in each 6-month interval of the postpartum year with ≥60 days between visits.

SECONDARY OUTCOMES:
Viral Suppression up to 1 year postpartum | Baseline through 1 year after delivery
  Viral Load ≤ 200 copies/mL using the last available Viral Load up to 180 days before the end of the postpartum year.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - MedStar Health Research Institute, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - Montefiore Medical Center/Albert Einstein College of Medicine, The Bronx, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Baylor College of Medicine, Houston, Texas